CLINICAL TRIAL: NCT02254122
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Inhalative Doses (20 µg, 50 µg, 100 µg, 200 µg and 400 µg) of BEA 2180 BR for 21 Days in Healthy Male Volunteers (Double-blind, Randomised, Placebo Controlled [at Each Dose Level] Study)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Inhalative Doses of BEA 2180 BR in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.2
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- BEA 2180 BR (Experimental)
  Interventions: Drug: BEA 2180 BR; Device: Respimat®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Respimat®

INTERVENTIONS:
Drug: BEA 2180 BR
  Arms: BEA 2180 BR
Drug: Placebo
  Arms: Placebo
Device: Respimat®

SUMMARY:
Study to investigate safety and tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of BEA 2180 BR

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria (examined at the Screening Visit):

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests

   1.1 No finding deviating from normal and of clinical relevance

   1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥30 and ≤55 years
3. BMI ≥18.5 and BMI < 30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. History of relevant orthostatic hypotension, fainting spells or blackouts
4. Chronic or relevant acute infections
5. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the Investigator
6. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
7. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
8. Participation in another trial with an investigational drug within two months prior to administration or during the trial
9. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
10. Inability to refrain from smoking during the trial
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range if indicative of underlying disease or poor health

Exclusion criteria specific for this study:

* Asthma or chronic obstructive pulmonary disease
* Glaucoma
* Urinary tract obstruction
* Occupational (professional) exposure to antimuscarinic substances

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2004-05; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to day 42
Number of subjects with clinically significant changes in vital signs | up to day 42
Number of subjects with clinically significant changes in 12-lead electrocardiogram | up to day 42
Number of subjects with clinically significant changes in laboratory parameters | up to day 42
Changes in effective airway resistance (Reff) | up to day 25
  Body plethysmography
Changes in specific effective airway conductance (SGeff) | up to day 25
  Body plethysmography
Changes in salivary secretion | up to day 21
Number of subjects with adverse events | up to day 42
Assessment of tolerability by the Investigator on a 4-point rating scale | day 42

SECONDARY OUTCOMES:
Maximum concentration of the analyte in plasma for several time points | up to day 35
Time from dosing to maximum concentration in plasma for several time points | up to day 35
Area under the concentration-time curve of the analyte in plasma for several time points | up to day 35
Amount of analyte that is eliminated in urine for several time points | up to day 34
Fraction of analyte excreted in urine for several time points | up to day 34
Renal clearance of the analyte in plasma for several time points | up to day 34
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval | up to day 35
Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose | up to day 35
Terminal rate constant in plasma at steady state (λz,ss) | up to day 35
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | up to day 35
Mean residence time of the analyte in the body after 21 administrations at steady state (MRTih,ss) | up to day 35
apparent clearance of the analyte in the plasma after extravascular administration at steady state (CL/F,ss) | up to day 35
apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state (Vz/F,ss) | up to day 35
Accumulation ratio (RA) of the analyte in plasma after multiple dose administration over a uniform dosing interval τ | up to day 35
Peak trough fluctuation (PTF) | up to day 35